CLINICAL TRIAL: NCT00603707
Title: Assessment of Whole Gut Transit Time Using the SmartPill Capsule: a Multi-Center Study
Brief Title: Assessment of Whole Gut Transit Time Using the SmartPill Capsule
Acronym: WholeGut
Status: Completed | Type: Observational
Sponsor: The SmartPill Corporation (Industry)
Responsible Party: John R. Semler/Chief Technology Officer, The SmartPill Corporation
Other Study IDs: 122205
Record Dates: First submitted 2008-01-08; First posted 2008-01-29 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Constipation
Keywords: capsule; constipation; whole gut transit; colonic transit; gastric emptying; small bowel transit
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: healthy adult subjects with no history or current gastrointestinal disorders or conditions
- Constipated: Adult subjects with functional constipation as define by Rome II criteria

SUMMARY:
Our null hypothesis states that the two techniques (Sitzmarks radioopaque markers and SmartPill) are equivalent and is demonstrated if the study population shows a correlation of 0.7 or higher.

DETAILED DESCRIPTION:
The purpose of the study is to measure total gastrointestinal transit time using SmartPill GI Monitoring System with pH.p Capsule and compare the transit time determined by capsule transit to the conventional radioopaque marker technique.

Both techniques are simultaneously applied in normal and constipated adult populations.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages of 18-80 years of age with functional constipation that fulfills the Rome II definition of functional constipation
* Bowel movement frequency of < 3 times per week but at least once per two weeks.
* Constipation symptoms for at least 1 year duration.
* Constipation, not abdominal pain, as the primary symptom.
* Ability to stop fiber, laxatives, prokinetic agents, and narcotic analgesic agents 3 days prior to the study and during the 5 day study period.
* Ability to stop proton pump inhibitors 7 days prior to the study and H2RAs for 3 days prior to the study.

Exclusion Criteria:

* Previous history of bezoars.
* Prior GI surgery except for cholecystectomy, appendectomy, or Nissen fundoplication
* Any abdominal surgery within the past 3 months
* Known or history of inflammatory bowel disease
* History of diverticulitis, diverticular stricture, and other intestinal strictures
* Tobacco use within eight hours prior to capsule ingestion and during the initial 8 hour recording on Day 0 or the Ingestion visit.
* Alcohol use within eight hours prior to capsule ingestion and throughout the entire monitoring period (5 days).
* BMI > 38
* Allergies to components of the SmartBar (Appendix IX).
* Females of childbearing age who are not practicing birth control and/or are pregnant or lactating. (A urine pregnancy test will be performed on female subjects prior to capsule ingestion).
* Cardiovascular, endocrine, renal, or other chronic disease likely to affect motility.
* Use of medical devices such as pacemakers, infusion pumps, or insulin pumps.
* Any contraindication to use of Fleets Enema or balloon expulsion test.
* Uncontrolled diabetes with a hemoglobin A1C greater than 10.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with constipation referred to a tertiary motility center
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
whole gut transit time | 2 days and 5 days

SECONDARY OUTCOMES:
Determine regional gut (gastric, small bowel, colonic) transit times | continuous time measure until caspule elimination

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Study Chair — Temple University Medical Center
Locations (8):
- United States (8):
  - Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - VA Medical Center, Buffalo, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Temple University Medical Center, Philadelphia, Pennsylvania